CLINICAL TRIAL: NCT04921345
Title: A Multicenter, Open-Label, Single-Group Clinical Trial to Assess the Pharmacokinetics, Safety and Efficacy of Nemolizumab (CD14152) in Pediatric Subjects (Aged 2 to 11 Years) With Moderate-to-Severe Atopic Dermatitis
Brief Title: Pharmacokinetics, Safety and Efficacy of Nemolizumab in Participants With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.118126
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Moderate-to-Severe Atopic Dermatitis
Keywords: Atopic Dermatitis; Nemolizumab; CD14152
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Participants aged 7-11 year (Experimental): Participants aged 7-11 years will receive nemolizumab for 52 weeks.
  Interventions: Drug: Nemolizumab
- Cohort 1.1: Participants aged 7-11 years (Experimental): Participants aged 7-11 years will receive nemolizumab for 52 weeks.
  Interventions: Drug: Nemolizumab
- Cohort 2: Participants aged 2-6 years (Experimental): Participants aged 2-6 years will receive nemolizumab for 52 weeks.
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Nemolizumab — Participants will receive subcutaneous (SC) injection of 10, 20 or 30 milligrams (mg) nemolizumab, every 4 weeks (Q4W) for 52 weeks with a loading dose of 20, 40 or 60 mg at Day 1 based on the body weight.
  Other Names: CD14152
  Arms: Cohort 1: Participants aged 7-11 year
Drug: Nemolizumab — Participants will receive SC injection of 5, 10 or 15 mg nemolizumab, Q4W for 52 weeks with a loading dose of 10, 20 or 30 mg at Day 1 based on the body weight.
  Other Names: CD14152
  Arms: Cohort 1.1: Participants aged 7-11 years; Cohort 2: Participants aged 2-6 years

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), efficacy, and safety of nemolizumab in pediatric participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic AD that has been documented for at least 6 months for participants aged 2-6 years and at least 1 year for participants aged 7-11 years before the screening visit and confirmed according to the American Academy of Dermatology Consensus Criteria at the time of the screening visit
* EASI score >=16 at both screening and baseline visits
* IGA score >=3 at both screening and baseline visits
* AD involvement >=10% of BSA at both screening and baseline visits
* Peak (maximum) PP NRS score of at least 4.0 at both screening and baseline visits
* Agree to apply a moisturizer throughout the study from the screening visit daily, and liberally as needed; agree to apply an authorized topical corticosteroids (TCS) from the screening visit and throughout the study as determined appropriate by the investigator
* Participant and caregiver willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Body weight less than 10 kilogram (kg)
* Child in Care: a child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation
* Participants with a current medical history of chronic bronchitis
* Requiring rescue therapy for AD during the run-in period or expected to require rescue therapy within 2 weeks following the baseline visit
* Positive serology results for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), hepatitis C (HCV) antibody with positive confirmatory test for HCV (example; polymerase chain reaction [PCR]), or human immunodeficiency virus (HIV) antibody at the screening visit
* History of lymphoproliferative disease, hypersensitivity (including anaphylaxis) to an immunoglobulin product and intolerance to low or mid potency topical corticosteroids
* Known or suspected immunosuppression
* Participants unwilling to refrain from using prohibited medications during the clinical trial.
* Other protocol defined exclusion criteria could apply

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Nemolizumab Serum Concentrations of Pediatric Participants | At Week 4, 8, 12, 16, 32 and 52
Apparent Total Body Clearance (Cl/F) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Apparent Volume of Distribution (Vd/F) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Absorption Rate Constant (Ka) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Maximum Observed Serum Concentration (Cmax) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Serum Concentration Observed Immediately Before Next Dosing (Ctrough) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Time to Reach the Maximum Observed Serum Concentration (Tmax) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Apparent Terminal Half-life (t1/2) of Nemolizumab | At Week 4, 8, 12, 16, 32 and 52
Number of Participants with Treatment Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESIs), Adverse Events Leading to Discontinuation and Serious Adverse Events (SAEs) | Baseline through Week 52

SECONDARY OUTCOMES:
Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis.
Number of Participants Achieving 50%, 75% or 90% Response From Baseline in Eczema Area and Severity Index (EASI-50, EASI-75 and EASI-90) at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  EASI assesses severity and extent of AD signs through a composite score of erythema, induration/population, excoriation, and lichenification. The severity will be assessed on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. The EASI score can range from 0 to 72 with higher scores representing greater severity of atopic dermatitis. EASI-50, EASI-75 and EASI-90 responders will be the participants who achieved >=50%, >=75% and >=90% overall improvement in EASI score respectively from baseline to Week 52.
Investigator's Global Assessment (IGA) Success Rate at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  IGA is a 5-point scale used by the investigator or trained designee to evaluate the global severity of AD. The Investigator will review the participant's skin and give a score of 0 (Clear), 1 (Almost clear), 2 (Mild), 3 (Moderate), or 4 (Severe).
Change From Baseline in Body Surface Area (BSA) Involvement by Atopic Dermatitis (AD) | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Absolute Change From Baseline in Weekly Average of Peak Pruritus Numeric Rating Scale (PP NRS) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Percent Change From Baseline in Weekly Average of Peak Pruritus Numeric Rating Scale (PP NRS) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Proportion of Participants With an Improvement of >= 4 From Baseline in Weekly Average of Peak Pruritus Numeric Rating Scale (PP NRS) at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Absolute Change From Baseline in Weekly Average of Average Pruritus Numeric Rating Scale (NRS) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Percent Change From Baseline in Weekly Average of Average Pruritus Numeric Rating Scale (NRS) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  Pruritus NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome.
Absolute Change From Baseline in Weekly Average of Sleep Disturbance Numeric Rating Scale (NRS) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants will be asked the following questions in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Higher scores indicate worse outcome.
Percent Change From Baseline in Weekly Average of Sleep Disturbance Numeric Rating Scale (NRS) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The sleep disturbance NRS is a scale used by the participants to report the degree of their sleep loss related to AD. Participants will be asked the following questions in their local language: how would you rate your sleep last night? On a scale of 0 to 10, with 0 being 'no sleep loss related to signs/symptoms of AD' and 10 being 'I cannot sleep at all due to the signs/symptoms of AD'. Higher scores indicate worse outcome.
Proportion of Participants Receiving any Rescue Therapy by Rescue Treatment | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score at Each Visit up to Week 52 | Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  SCORAD is a clinical tool for assessing the severity and the extent of AD signs and symptoms. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Change From Baseline in Children's Dermatology Life Quality Index (cDLQI) For Participants >=4 Years of Age up to Week 16 and Week 52 | Baseline, Week 16 and Week 52
  The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily activities, leisure, work/school, personal relationships, and treatment. The participant will rate each question ranging from 0 (not at all) to 3 (very much) and score ranges from 0 to 30. A higher total score indicates a poorer quality of life (QoL).
Change From Baseline in Infants' Dermatology Life Quality Index (iDLQI) For Participants <4 Years of Age From Baseline up to Week 16 and up to Week 52 | Baseline, Week 16 and Week 52
  The DLQI is a validated 10-item questionnaire covering domains including symptoms/feelings, daily activities, leisure, work/school, personal relationships, and treatment. The participant will rate each question ranging from 0 (not at all) to 3 (very much) and score ranges from 0 to 30. A higher total score indicates a poorer quality of life (QoL).
Change From Baseline in Patient-Oriented Eczema Measure (POEM) up to Week 16 and Week 52 | Baseline, Week 16 and Week 52
  The POEM is a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Pharmacokinetic (PK)/Pharmacodynamic (PD) Relationship Between Nemolizumab Serum Concentration and Changes in Peak Pruritus Numeric Rating Scale (PP NRS) | Baseline, Week 16 and Week 52
  The relationship between nemolizumab serum concentrations will be evaluated using correlation and/or linear regression methods to evaluate possible associations with changes in PP-NRS score.
Pharmacokinetic (PK)/Pharmacodynamic (PD) Relationship Between Nemolizumab Serum Concentration and Changes in Eczema Area and Severity Index (EASI) Score | Baseline, Week 16 and Week 52
  The relationship between nemolizumab serum concentrations will be evaluated using correlation and/or linear regression methods to evaluate possible associations with changes in EASI score.
Pharmacokinetic (PK)/Pharmacodynamic (PD) Relationship Between Nemolizumab Serum Concentration and Changes in Investigator's Global Assessment (IGA) Score | Baseline, Week 16 and Week 52
  The relationship between nemolizumab serum concentrations will be evaluated using correlation and/or linear regression methods to evaluate possible associations with changes in IGA score.
Number of Participants with Positive Anti-Drug Antibody (ADA) for Nemolizumab | Baseline, Week 16 and Week 52

CONTACTS AND LOCATIONS:
Locations (23):
- United States (14):
  - Galderma Investigational Site #8636, Fountain Valley, California
  - Galderma Investigational Site #9937, San Diego, California
  - Galderma Investigational Site #9930, Vista, California
  - Galderma Investigational Site #9929, Coral Gables, Florida
  - Galderma Investigational Site #8142, Indianapolis, Indiana
  - Galderma Investigational Site #8092, Louisville, Kentucky
  - Galderma Investigational Site #8155, Troy, Michigan
  - Galderma Investigational Site #8560, West Bloomfield, Michigan
  - Galderma Investigational Site #8242, Brooklyn, New York
  - Galderma Investigational Site #9938, New York, New York
  - Galderma Investigational Site #8206, Norman, Oklahoma
  - Galderma Investigational Site #8255, Philadelphia, Pennsylvania
  - Galderma Investigational Site #9931, Beaumont, Texas
  - Galderma Investigational Site #78218-3128, San Antonio, Texas
- Galderma Investigational Site #6218, Hellerup, Denmark
- Hungary (2):
  - Galderma Investigational Site #6147, Budapest
  - Galderma Investigational Site #5531, Szeged
- Poland (5):
  - Galderma Investigational Site #5570, Lodz
  - Galderma Investigational Site #6237, Ostrowiec Świętokrzyski
  - Galderma Investigational Site #5495, Rzeszów
  - Galderma Investigational Site #6262, Warsaw
  - Galderma Investigational Site #6261, Wroclaw
- Galderma Investigational Site #5896, Esplugues de Llobregat, Spain